CLINICAL TRIAL: NCT02600013
Title: Locomotor Training With the Exoskeleton EKSO-GT in Patients With Incomplete Motor Spinal Cord Injury in a Hospital Setting: an Observational Study
Brief Title: Locomotor Training With Exoskeleton EKSO-GT in Patients With Incomplete Motor Spinal Cord Injury in a Hospital Setting
Status: Completed | Type: Observational
Sponsor: Montecatone Rehabilitation Institute S.p.A. (Other)
Responsible Party: Sponsor
Other Study IDs: CE-15093
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Spinal Cord Injuries
Keywords: incomplete motor SCI; robotic gait training; exoskeleton; rehabilitation tool; EKSO-GT
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this observational, non-controlled, non-profit study is to describe the responses to rehabilitative training with the robotic exoskeleton EKSO-GT in patients with incomplete motor Spinal Cord Injury (AIS C or D). Such rehabilitative tool is employed during inpatient intensive rehabilitation in a 3rd level Italian hospital. Safety and tolerability of the device are also assessed and described.

DETAILED DESCRIPTION:
The locomotor training, defined as any "therapeutic program aimed at the recovery of walking through intense practice of the task of walking", is a very important part of the treatment plan for patients with locomotor dysfunction of the lower extremities and is aimed at retraining the nervous system, facilitating the recovery of muscle strength, improving balance and voluntary motor coordination. In fact, the majority of gait rehabilitation strategies is based on the concept of plasticity of the Central Nervous System and of "Central Pattern Generator": this plasticity is supposed to be facilitated by early, intensive and specific therapies, able to enhance the natural recovery processes.

The final goal is to help patients regain the highest level of personal autonomy which consequently translates also in a better overall quality of life.

The anthropomorphic robotic exoskeleton EKSO (Ekso Bionics, USA) is designed to assist in upright, weight bearing over ground gait training of people with weakness or paralysis of the lower limbs, due to a disorder, a disease or a neurologic injury. The training with EKSO is possible even in the presence of minimal forearm strength in order to resting to an upfront mobile walker. The device is available on the market for some years and it has recently been introduced in the clinical practice of some Italian rehabilitative centers. Montecatone Rehabilitation Institute acquired the most recent "GT" version of EKSO that enables variable, adaptive assistance.

This observational, longitudinal research study has a descriptive/exploratory intent. It aims at describing the responses to rehabilitative training with the robotic exoskeleton EKSO-GT in a cohort of incomplete motor Spinal Cord Injury patients (AIS C or D), as a rehabilitative tool in a setting of intensive inpatient rehabilitation (3rd level hospital). Safety and tolerability are also assessed and described.

This kind of study is justified by the fact that although the global network of professional users agree on the potential of such "young" technology on rehabilitation outcomes, few are the clinical data published in the scientific literature in relation to its use. It is believed that the results obtained from this study will be useful for the future definition of better protocols of use of the exoskeleton, more specific for the different types of SCI people.

Primary objective: to describe the responses to the robotic over ground gait training with EKSO-GT in an inpatient rehabilitative hospital setting, in people with incomplete motor SCI (AIS C or D). This objective is achieved by means of the administration of walking tests and the assessment of both lower limbs motor function and kinetic and endurance characteristics of walking.

Secondary objectives, description in the same patients' population:

* Safety and tolerability of locomotor training with the EKSO-GT;
* Level of strength and muscle trophism of the patient subjected to the robotic training;
* Any reductions in pain and/or spasticity due to SCI during and after the locomotor training with the EKSO-GT;
* Quality of life and mood status of patients;
* Level of patient satisfaction in relation to the gait training with the EKSO-GT;
* Maintenance of any acquired benefits (follow-up 45 days after the conclusion of the training with the EKSO-GT), with respect to most outcomes taken into account.

All functional assessments are carried out when the patient does not wear the exoskeleton; however, functional gait specific test (10-meter walk test and 6-minutes walk test) are performed when the exoskeleton is worn and when it is not worn only by those patients able to accomplish those gait specific tests in such a way.

For gait specific tests the first evaluation with the exoskeleton worn is programmed to the third robotic rehabilitative session, as the first sessions are necessary for set-up purposes.

Data on the safety and tolerability of the EKSO-GT training are recorded at the beginning and at the end of each session, however a synthesis of safety outcomes will be carried out at predefine time frames.

The training with the EKSO-GT is carried out in addition to the "conventional" locomotor training and in the presence of specifically trained physiotherapists, always under medical supervision.

Patients undergo 12 or 18 rehabilitative EKSO sessions, 2-3 times per week, of max 1 hr each.

ELIGIBILITY:
Inclusion Criteria:

* inpatient consecutive SCI subjects;
* incomplete motor SCI of any etiology, classified as AIS C or D;
* ability to rest the upper limbs on a mobile support (e.g. walker);
* orthostatic exercise well tolerated for at least 60 continuously minutes and regularly exercised; or regular locomotor exercise; or ability of functional walk;
* sufficient range of motion (ROM) of lower limbs joints to achieve a mutual path pattern and allow transition from sitting to vertical position;
* height: minimum 157 cm, maximum 188 cm;
* maximum weight: 100 kg;
* intertrochanteric maximum distance: 46 cm;
* stable medical condition;
* intact cognitive abilities and full cooperation of the subject;
* research informed consent signed.

Exclusion Criteria:

* skin lesions in areas of EKSO contact;
* instability or major deformity of the spine;
* limbs joint instability;
* indication to the use of spinal orthoses;
* presence of uncontrolled spasticity (score > 3 of the Modified Ashworth Scale) in most of the muscle groups of the lower limbs;
* active acute deep vein thrombosis;
* uncontrolled, severe and recurrent autonomic dysreflexia;
* significant bone fragility;
* recent traumatic and/or pathological bone fractures, significant for the required training;
* limb-length discrepancy for femur length (> 1.3 cm) and leg length (> 1.9 cm);
* neurogenic paraosteoarthropathy (at onset or inflammatory);
* symptomatic orthostatic hypotension;
* cardiopulmonary comorbidities limiting exertion;
* documented psychiatric condition that might hinder the training with EKSO-GT;
* active pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incomplete motor SCI patients in a setting of inpatient intensive rehabilitation (3rd level hospital)
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in 10-Meter walk test with EKSO worn | baseline (session 3, up to 1 week), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks)
Change in 6-Minutes walk test with EKSO worn | baseline (session 3, up to 1 week), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks)
Change in 10-Meter walk test with EKSO not worn (if able) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks)
Change in 6-Minutes walk test with EKSO not worn (if able) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks)

SECONDARY OUTCOMES:
Change in 10-Meter walk test | Follow-up: 45 days after EKSO training closing session 12 or 18
  Possible only on those patients able to perform the test without wearing the EKSO during the rehabilitative sessions
Change in 6-Minutes walk test | Follow-up: 45 days after EKSO training closing session (12 or 18)
  Possible only on those patients able to perform the test without wearing the EKSO during the rehabilitative sessions
Change in score of the Walking Index for Spinal Cord Injury, version II (WISCI-II) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change in score of the Mobility part of the Spinal Cord Independence Measure scale, version III (SCIM III) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change in number of footsteps made when EKSO is worn and actual locomotion is in place | Immediately after the end of each rehabilitative session
  Although measurements are taken on each rehabilitative session, an overall evaluation is carried out also at: baseline (session 3, up to 1 week), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Change in actual locomotion time when EKSO is worn | Immediately after the end of each rehabilitative session
  Although measurements are taken on each rehabilitative session, an overall evaluation is carried out also at: baseline (session 3, up to 1 week), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks). This measurement is needed to standardize the progression in walking of each patient, when the EKSO is worn. The formula of the combined, standardized outcome is: "Number of footsteps made when EKSO is worn and actual locomotion is in place" divided by "Actual locomotion time when EKSO is worn"
Change in blood pressure during EKSO rehabilitative sessions | Immediately before the beginning of each EKSO rehabilitative session, immediately after the end of each EKSO rehabilitative session
  This outcome covers a safety issue and for this reason measurements are taken on each rehabilitative session. However, an overall evaluation is carried out also at: baseline (initial visit), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Change in heart rate during EKSO rehabilitative sessions | Immediately before the beginning of each EKSO rehabilitative session, immediately after the end of each EKSO rehabilitative session
  This outcome covers a safety issue and for this reason measurements are taken on each rehabilitative session. However, an overall evaluation is carried out also at: baseline (initial visit), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Change in peripheral O2 saturation during each EKSO rehabilitative session | Immediately before the beginning of each EKSO rehabilitative session, immediately after the end of each EKSO rehabilitative session
  This outcome covers a safety issue and for this reason measurements are taken on each rehabilitative session. However, an overall evaluation is carried out also at: baseline (initial visit), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Number of falls during the whole rehabilitation period with EKSO (worn) | Immediately before the beginning of each EKSO rehabilitative session, immediately after the end of each EKSO rehabilitative session
  This outcome covers a safety issue and for this reason measurements are taken on each rehabilitative session. However, an overall evaluation is carried out also at: baseline (initial visit), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Onset of pain due to EKSO wearing (NRS scale) | Immediately before the beginning of each EKSO rehabilitative session, immediately after the end of each EKSO rehabilitative session
  This outcome covers a safety issue and for this reason measurements are taken on each rehabilitative session. However, an overall evaluation is carried out also at: baseline (initial visit), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Onset of pressure ulcers due to EKSO wearing | Immediately before the beginning of each EKSO rehabilitative session, immediately after the end of each EKSO rehabilitative session
  This outcome covers a safety issue and for this reason measurements are taken on each rehabilitative session. However, an overall evaluation is carried out also at: baseline (initial visit), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Classification of any pressure ulcers emerged due to EKSO wearing, according to the international classification of the European and US National Pressure Ulcer Advisory panels (EPUAP and NPUAP), along with the Pan Pacific Pressure Injury Alliance (PPPIA) | Immediately before the beginning of each EKSO rehabilitative session, immediately after the end of each EKSO rehabilitative session
  This outcome covers a safety issue and for this reason measurements are taken on each rehabilitative session. However, an overall evaluation is carried out also at: baseline (initial visit), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Onset of musculoskeletal complications due to EKSO rehabilitation | Immediately before the beginning of each EKSO rehabilitative session, immediately after the end of each EKSO rehabilitative session
  This outcome covers a safety issue and for this reason measurements are taken on each rehabilitative session. However, an overall evaluation is carried out also at: baseline (initial visit), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Onset of other complications due to EKSO rehabilitation | Immediately before the beginning of each EKSO rehabilitative session, immediately after the end of each EKSO rehabilitative session
  This outcome covers a safety issue and for this reason measurements are taken on each rehabilitative session. However, an overall evaluation is carried out also at: baseline (initial visit), session 12 (up to 6 weeks) and session 18 if any (up to 9 weeks)
Change in spasticity (Modified Ashworth Scale) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change in pain (ISCI Pain Basic Data Set) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change in limbs muscular strength: Total ASIA Lower Extremity Motor Score (LEMS) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change in limbs muscular strength: Partial ASIA LEMS score "Lower Extremity Right" (LER) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change in limbs muscular strength: Partial ASIA LEMS score "Lower Extremity Left" (LEL) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change in lower limbs muscular trophism (circumference of right thigh) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change in lower limbs muscular trophism (circumference of left thigh) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change of rehabilitative potential: 100 minus the actual Spinal Cord Injury Ability Realization Measurement Index (SCI-ARMI) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change of quality of life (ISCI Quality of Life Basic Data Set) | Baseline (initial visit), session 12 (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Change of mood status (POMS questionnaire) | Baseline (initial visit), session 12 if end of training (up to 6 weeks), session 18 if any (up to 9 weeks), 45 days after EKSO training closing session
Level of patient satisfaction in the use of the EKSO (ad hoc questionnaire) | Last EKSO training session (up to 9 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jacopo Bonavita, Dir Spinal U, Principal Investigator — Montecatone Rehabilitation Institute S.p.A.
Locations (1):
- Montecatone Rehabilitation Institute S.p.A., Imola, BO, Italy